CLINICAL TRIAL: NCT06048900
Title: Evaluation of the Effect of Trendelenburg Position Time on Intracranial Pressure in Laparoscopic With Ultrasonographic Optic Nerve Sheath Diameter Measurement
Brief Title: Evaluation of the Effect of Trendelenburg Position Duration on Intracranial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek Cetinkaya (Other)
Responsible Party: Sponsor-Investigator, Dilek Cetinkaya, Associate Professor, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ESOGU1
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Intracranial Pressure Increase
Keywords: optic nerve sheath diameter measurement; trendelenburg position; laparoscopic hysterectomy
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: In patients in head-down position who will undergo laparoscopic hysterectomy, it is planned to measure the optic nerve sheath diameter with ultrasound at the beginning and at certain periods of the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optic nerve sheath diameter measurements (Other): A total of 7 measurements were planned to be made at specified times.
  Interventions: Device: ultrasound guided optic nerve sheath diameter measurement

INTERVENTIONS:
Device: ultrasound guided optic nerve sheath diameter measurement — First, both eyes were measured in a neutral position while awake and after intubation. Measurements were made at regular intervals until the end of the operation after the head-down position and in the neutral position after the operation.

SUMMARY:
The Lloyd Davies position is a position used in laparoscopic hysterectomies where the head is lowered 45 degrees and the legs are bent from the knee area.It is a version of the Trendelenburg position. Both this position and for laparoscopic surgery carbon dioxide (CO2) gas given into the abdomen, causes problems for the patient. Increased abdominal and thoracic pressure impairs venous return and increases intracranial pressure. Optic nerve sheath diameter can be measured by placing an ultrasound probe over the eye. It is possible to follow up the increase in intracranial pressure with this diameter measurement. In this study, it was planned to measure the optic nerve sheath diameter by ultrasound in patients who will undergo laparoscopic hysterectomy. It is aimed to observe the changes in the increase in intracranial pressure as the time lengthens with the measurements to be made at certain intervals during the operation. Secondary aim is to determine whether there is a cut-off value where the intracranial pressure starts to increase.

DETAILED DESCRIPTION:
The Trendelenburg position is the patient's head down with the table tilted, with the head closer to the floor than the feet. Lloyd Davies position is a modified version of the Trendelenburg position, used especially in laparoscopic hysterectomies, where the head is lowered 30-45° and the legs are bent at knee level. During this surgery, pneumoperitoneum is also applied by administering carbon dioxide (CO2) into the abdomen. During this surgery, pneumoperitoneum is also applied by administering CO2 into the abdomen. The applied position and intra-abdominal CO2 cause some physiological changes. These changes include respiratory and cardiac changes as well as increased intracranial pressure. Optic nerve sheath diameter can be measured by placing an ultrasound probe over the eye. Increase in intracranial pressure can be followed by sequential measurements. In this study, it was planned to measure the optic nerve sheath diameter by ultrasound in patients who will undergo laparoscopic hysterectomy. It is aimed to observe the changes in the increase in intracranial pressure as the time lengthens with the measurements to be made at certain intervals during the operation. Before the patients were given anesthesia induction, optic nerve sheath diameter measurement (ONSD) was performed by imaging in the sagittal and transverse planes in both eyes in neutral position. The second measurement was taken 2 minutes after endotracheal intubation in the neutral position. After the trocars were placed and pneumoperitoneum was applied, the patient was placed in the Lloyd Davies position. After the position was given, bilateral ONSD measurements were taken at the 30th minute, 60th minute, 75th minute, and 90th minute. At the end of the surgery, pneumoperitoneum and position were neutralized. The last measurement was taken 5 minutes after the patient was placed in the neutral position. Near infrared spectrometry (NIRS) monitoring was performed throughout the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo laparoscopic hysterectomy

Exclusion Criteria:

* chronic lung disease, pulmonary hypertension
* glaucoma
* history of eye surgery
* diabetic retinopathy
* intracranial mass,
* hydrocephalus
* history of intracranial surgery
* American society of anesthesiology (ASA) physical classification IV
* optic neuritis
* who do not want to participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients who will undergo laparoscopic hysterectomy
Enrollment: 25 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter measurement | during the surgery
  increase in optic nerve sheath diameter

SECONDARY OUTCOMES:
Timing of increased intracranial pressure | during the surgery
  If the sheath diameter is over 5 mm, increased pressure will be accepted.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Çetinkaya, Study Chair — Eskisehir Osmangazi University Medical Faculty
Locations (1):
- Eskisehir Osmangazi University Medical Faculty, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Chin JH, Seo H, Lee EH, Lee J, Hong JH, Hwang JH, Kim YK. Sonographic optic nerve sheath diameter as a surrogate measure for intracranial pressure in anesthetized patients in the Trendelenburg position. BMC Anesthesiol. 2015 Mar 31;15:43. doi: 10.1186/s12871-015-0025-9. eCollection 2015. PMID 25861241
- [Background] Ohle R, McIsaac SM, Woo MY, Perry JJ. Sonography of the Optic Nerve Sheath Diameter for Detection of Raised Intracranial Pressure Compared to Computed Tomography: A Systematic Review and Meta-analysis. J Ultrasound Med. 2015 Jul;34(7):1285-94. doi: 10.7863/ultra.34.7.1285. PMID 26112632
- [Derived] Guloglu H, Cetinkaya D, Oge T, Bilir A. Evaluation of the effect of trendelenburg position duration on intracranial pressure in laparoscopic hysterectomies using ultrasonographic optic nerve sheath diameter measurements. BMC Anesthesiol. 2024 Jul 15;24(1):238. doi: 10.1186/s12871-024-02624-4. PMID 39010013